CLINICAL TRIAL: NCT00689377
Title: Prevalence of Peripheral Arterial Disease in Subjects With a Moderate CVD Risk, With No Overt Vascular Diseases nOR diAbetes Mellitus
Brief Title: Prevalence of Peripheral Arterial Disease in Subject With a Moderate Risk of Cardiovascular (CV) Disease (CVD) in Primary Prevention
Acronym: PANDORA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CEU-DUM-2006/1
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Peripheral Arterial Disease (PAD); Moderate Risk for Cardiovascular Disease (CVD)
Keywords: Peripheral Arterial Disease (PAD); Cardiovascular Disease (CVD); Atherosclerotic cardiovascular disease; Atherosclerosis; Primary CVD prevention
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Subjects of either sex, any race, with at least two CVD risk factors, with no overt cardiovascular diseases nor diabetes mellitus

SUMMARY:
Non interventional study aimed to establish the prevalence of lower extremity peripheral arterial disease (PAD), defined as an ankle-brachial index (ABI) not above 0.90 in subjects with a moderate risk of cardiovascular disease, with no overt cardiovascular diseases nor diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male subject aged 45 years or above, or female subject aged 55 years or above (age-related CVD risk factor)
* At least another of the following risk factor for CVD: cigarette smoking, hypertension, low HDL cholesterol or high LDL cholesterol, family history of premature coronary heart disease, elevated waist circumference
* Willingness to participate in the survey and complying with the study by signing a written informed consent

Exclusion Criteria:

* No or 1 risk factor for CVD; symptoms of PAD; diabetes mellitus; coronary heart disease or equivalents
* No lipid data collected in the last 12 months
* Serious or unstable medical or psychological conditions that, in the opinion of the Investigator, would compromise the subject's safety or successful participation in the study; unwilling or unable to provide informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of either sex, any race, with at least two CVD risk factors, with no overt cardiovascular diseases nor diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of lower extremities peripheral arterial disease (PAD), in subjects with a moderate CVD risk, with no overt cardiovascular diseases nor diabetes mellitus | 1 visit

SECONDARY OUTCOMES:
Prevalence of cardiovascular risk factors in subjects with at least two CVD risk factors, with no overt cardiovascular diseases nor diabetes mellitus | 1 visit
Cardiovascular risk level and risk factor treatment in the selected population assessed according to the locally adopted risk charts or algorithms | 1 visit
Determinants (i.e., subject and physician characteristics) for PAD underdiagnosis in the selected population | 1 visit

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Sabia, Study Director — AstraZeneca S.p.A.; Mario Mangrella, Study Chair — AstraZeneca S.p.A; Claudio Cimminiello, Study Chair — Unit of Medicine, Vimercate Hospital - Vimercate (MI) - Italy; Claudio Borghi, Study Chair — Internal Medicine Dept., di Medicina Interna, Policlinico Universitario Sant'Orsola-Malpighi, Bologna, Italy
Locations (331):
- Belgium (103):
  - Research Site, Chênée, Liege
  - Research Site, Aarschot
  - Research Site, Alsemberg
  - Research Site, Anderlecht
  - Research Site, Anthée
  - Research Site, Arendonk
  - Research Site, Assenede
  - Research Site, Baisy-Thy
  - Research Site, Bande
  - Research Site, Beringen
  - Research Site, Bertrix
  - Research Site, Beyne-Heusay
  - Research Site, Biesme-sous-Thuin
  - Research Site, Brussels
  - Research Site, Burdinne
  - Research Site, Cerexhe-Heuseux
  - Research Site, Champion
  - Research Site, De Pinte
  - Research Site, Deurle
  - Research Site, Dolembreux
  - Research Site, Dottignies
  - Research Site, Dour
  - Research Site, Drongen
  - Research Site, Ecaussinnes
  - Research Site, Eeklo
  - Research Site, Eisden
  - Research Site, Eke-Nazareth
  - Research Site, Ekeren
  - Research Site, Ellezelles
  - Research Site, Evergem
  - Research Site, Feluy
  - Research Site, Fléron
  - Research Site, Forest
  - Research Site, Fosses-la-Ville
  - Research Site, Geel
  - Research Site, Gent (Sint-Amandsberg)
  - Research Site, Ghent
  - Research Site, Gilly
  - Research Site, Gozée
  - Research Site, Grez-Doiceau
  - Research Site, Gribomont
  - Research Site, Ham
  - Research Site, Hasselt
  - Research Site, Hoboken
  - Research Site, Hooglede
  - Research Site, Koekelberg (Brussl)
  - Research Site, Koksijde
  - Research Site, Kraainem
  - Research Site, Landelies
  - Research Site, Ledeberg (Gent)
  - Research Site, Leopoldsburg
  - Research Site, Lillois
  - Research Site, Linkebeek
  - Research Site, Lommel
  - Research Site, Lustin
  - Research Site, Maasmechelen
  - Research Site, Malmedy
  - Research Site, Marchienne-au-Pont
  - Research Site, Marchovelette
  - Research Site, Melsbroek
  - Research Site, Mettet
  - Research Site, Molenbeek
  - Research Site, Molenbeek-Saint-Jean
  - Research Site, Natoye
  - Research Site, Oosteeklo
  - Research Site, Oostham
  - Research Site, Oud-Turnhout
  - Research Site, Oudenaarde
  - Research Site, Quaregnon
  - Research Site, Rance
  - Research Site, Ransart
  - Research Site, Retie
  - Research Site, Rode
  - Research Site, Ronquières
  - Research Site, Rosières
  - Research Site, Scherpenheuvel
  - Research Site, Seraing
  - Research Site, Sint-Agatha-Rode
  - Research Site, Sint-Amandsberg
  - Research Site, Sint-Denijs-Westrem
  - Research Site, Sint-Martens-Latem
  - Research Site, Spouwen
  - Research Site, Sprimont
  - Research Site, Steenokkerzeel
  - Research Site, Tessenderlo
  - Research Site, Thuillies
  - Research Site, Thuin
  - Research Site, Tielt
  - Research Site, Turnhout
  - Research Site, Uccle
  - Research Site, Velroux
  - Research Site, Veurne
  - Research Site, Vlimmeren
  - Research Site, Vosselaar
  - Research Site, Waarschoot
  - Research Site, Waremme
  - Research Site, Waterloo
  - Research Site, Weelde
  - Research Site, Wellin
  - Research Site, Wetteren
  - Research Site, Wezembeek
  - Research Site, Willebroek
  - Research Site, Zomergem
- France (92):
  - Research Site, Agde
  - Research Site, Antony
  - Research Site, Arsac
  - Research Site, Aubervilliers
  - Research Site, Baho
  - Research Site, Balma
  - Research Site, Beauzelle
  - Research Site, Bérat
  - Research Site, Béziers
  - Research Site, Blois
  - Research Site, Bourg-la-Reine
  - Research Site, Bourg-lès-Valence
  - Research Site, Carnon-Plage
  - Research Site, Carquefou
  - Research Site, Castets
  - Research Site, Champforgeuil
  - Research Site, Champigny-sur-Marne
  - Research Site, Chatillon Coumont
  - Research Site, Collioure
  - Research Site, Colomiers
  - Research Site, Courpière
  - Research Site, Cremeaux
  - Research Site, Derval
  - Research Site, Domène
  - Research Site, Drancy
  - Research Site, Eyragues
  - Research Site, Fontaine
  - Research Site, Fresnes-sur-Escaut
  - Research Site, Gargenville
  - Research Site, Garons
  - Research Site, Goven
  - Research Site, Guérande
  - Research Site, Herbignac
  - Research Site, Houilles
  - Research Site, Hyères
  - Research Site, Issy-les-Moulineaux
  - Research Site, Ivry-sur-Seine
  - Research Site, La Baule-Escoublac
  - Research Site, La Courneuve
  - Research Site, La Riche
  - Research Site, Lattes
  - Research Site, Le Coudray-Montceaux
  - Research Site, Le Temple-de-Bretagne
  - Research Site, Lembach
  - Research Site, Longages
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Martigues
  - Research Site, Metz
  - Research Site, Meylan
  - Research Site, Mezel
  - Research Site, Mirabeau
  - Research Site, Montigny-lès-Metz
  - Research Site, Montpellier
  - Research Site, Mouchin
  - Research Site, Mouvaux
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Noisy-le-Grand
  - Research Site, Oignies
  - Research Site, Orliénas
  - Research Site, Paris
  - Research Site, Pauillac
  - Research Site, Pernes-les-Fontaines
  - Research Site, Pérols
  - Research Site, Plan-de-Cuques
  - Research Site, Pontcharra
  - Research Site, Rieumes
  - Research Site, Ris-Orangis
  - Research Site, Roanne
  - Research Site, Rosny-sous-Bois
  - Research Site, Saint Donat L Herbasse
  - Research Site, Saint-Etienne
  - Research Site, Saint-Galmier
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Ouen
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Sébastien-de-Morsent
  - Research Site, Sauveterre-de-Guyenne
  - Research Site, Seraincourt
  - Research Site, Tarascon
  - Research Site, Thizy
  - Research Site, Toulon
  - Research Site, Tours
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villenave-d'Ornon
  - Research Site, Villette-d'Anthon
  - Research Site, Villeurbanne
  - Research Site, Villé
  - Research Site, Vincennes
  - Research Site, Wittelsheim
- Greece (50):
  - Research Site, Agrinio
  - Research Site, Alexandroupoli
  - Research Site, Arta
  - Research Site, Athens
  - Research Site, Athens North 1
  - Research Site, Attika South
  - Research Site, Attiki
  - Research Site, Chalkidiki
  - Research Site, Chania
  - Research Site, Chrisoupoli Kavalas
  - Research Site, Corfu
  - Research Site, Corinth
  - Research Site, Drama
  - Research Site, Giannitsá
  - Research Site, Ioannina
  - Research Site, Iraklio Kritis
  - Research Site, Itháki
  - Research Site, Kalamaria
  - Research Site, Kalamata
  - Research Site, Karpenisi
  - Research Site, Kastoria
  - Research Site, Katerini
  - Research Site, Kavala
  - Research Site, Kilkis
  - Research Site, Komotini
  - Research Site, Koropí
  - Research Site, Kozani
  - Research Site, Lakonia
  - Research Site, Lamia
  - Research Site, Larissa
  - Research Site, Nafpaktos
  - Research Site, Pátrai
  - Research Site, Pírgos
  - Research Site, Ptolemaida
  - Research Site, Rest of Salonica
  - Research Site, Rethymno
  - Research Site, Rhodes
  - Research Site, Salonica Central East
  - Research Site, Salonica Central West
  - Research Site, Salonica Suburbs East
  - Research Site, Salonica Suburbs West
  - Research Site, Serres
  - Research Site, Sitia Kritis
  - Research Site, Trikala
  - Research Site, Tripoli
  - Research Site, Véria
  - Research Site, Volos
  - Research Site, Xalkida
  - Research Site, Xánthi
  - Research Site, Zakynthos
- Italy (23):
  - Research Site, AL
  - Research Site, AR
  - Research Site, AT
  - Research Site, BA
  - Research Site, Bò
  - Research Site, CE
  - Research Site, CO
  - Research Site, FI
  - Research Site, FR
  - Research Site, GR
  - Research Site, MI
  - Research Site, MN
  - Research Site, NU
  - Research Site, OG
  - Research Site, OR
  - Research Site, PE
  - Research Site, RC
  - Research Site, SA
  - Research Site, SR
  - Research Site, TO
  - Research Site, TP
  - Research Site, VI
  - Research Site, VT
- Netherlands (31):
  - Research Site, 's-Hertogenbosch
  - Research Site, Beek en Donk
  - Research Site, Beerzerveld
  - Research Site, Bennebroek
  - Research Site, Berlicum
  - Research Site, Deurne
  - Research Site, Dordrecht
  - Research Site, Echt
  - Research Site, Ermelo
  - Research Site, Hengelo
  - Research Site, Hoogwoud
  - Research Site, Huizen
  - Research Site, Hulst
  - Research Site, Landgraaf
  - Research Site, Lichtenvoorde
  - Research Site, Lieshout
  - Research Site, Lisse
  - Research Site, Losser
  - Research Site, Nijmegen
  - Research Site, Oude Pekela
  - Research Site, Poortvliet
  - Research Site, Rijswijk
  - Research Site, Roelofarendsveen
  - Research Site, Rotterdam
  - Research Site, Sgravenzande
  - Research Site, Soerendonk
  - Research Site, Spijkenisse
  - Research Site, The Hague
  - Research Site, Wassenaar
  - Research Site, Wildervank
  - Research Site, Woerden
- Switzerland (32):
  - Research Site, Allschwil
  - Research Site, Balerna
  - Research Site, Basel
  - Research Site, Bellinzona
  - Research Site, Brittnau
  - Research Site, Bülach
  - Research Site, Camorino
  - Research Site, Chiasso
  - Research Site, Claro
  - Research Site, Coldrerio
  - Research Site, Dallikon
  - Research Site, Dornach
  - Research Site, Düdingen
  - Research Site, La Tour-de-Peilz
  - Research Site, Laufenburg
  - Research Site, Lausanne
  - Research Site, Lugano
  - Research Site, Melide
  - Research Site, Monthey
  - Research Site, Muttenz
  - Research Site, Ponte Capriasca
  - Research Site, Reinach
  - Research Site, Renens VD
  - Research Site, Rümlang
  - Research Site, St-Maurice
  - Research Site, Stabio
  - Research Site, Stäfa
  - Research Site, Tesserete
  - Research Site, Thalwil
  - Research Site, Vevey
  - Research Site, Winterthur
  - Research Site, Zurich

REFERENCES:
- [Derived] Sanna G, Alesso D, Mediati M, Cimminiello C, Borghi C, Fazzari AL, Mangrella M; PANDORA study investigators. Prevalence of peripheral arterial disease in subjects with moderate cardiovascular risk: Italian results from the PANDORA study Data from PANDORA (Prevalence of peripheral Arterial disease in subjects with moderate CVD risk, with No overt vascular Diseases nor Diabetes mellitus). BMC Cardiovasc Disord. 2011 Oct 7;11:59. doi: 10.1186/1471-2261-11-59. PMID 21981988
- [Derived] Cimminiello C, Borghi C, Kownator S, Wautrecht JC, Carvounis CP, Kranendonk SE, Kindler B, Mangrella M; PANDORA Study Investigators. Prevalence of peripheral arterial disease in patients at non-high cardiovascular risk. Rationale and design of the PANDORA study. BMC Cardiovasc Disord. 2010 Aug 5;10:35. doi: 10.1186/1471-2261-10-35. PMID 20687927